CLINICAL TRIAL: NCT00696956
Title: Paclitaxel Coated Balloons for Prevention of Restenosis in Small Arteries Below the Knee Compared to Angioplasty Using Uncoated Balloons
Brief Title: Drug Coated Balloons for Prevention of Restenosis
Acronym: Piccolo
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital Tuebingen (Other)
Responsible Party: Prof. Dr. med. Gunnar Tepe, Universtiy of Tuebingen
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Pac-3; Pac-3
Record Dates: First submitted 2008-06-10; First posted 2008-06-13 (Estimated); Last update posted 2008-06-13 (Estimated); Status verified 2008-05

CONDITIONS: Atherosclerosis; Restenosis; Limb Ishemia
Keywords: local drug delivery; balloon angioplasty; safety and tolerance of paclitaxel coated PTA balloons; in inhibiting restenosis of below the knee arteries; Efficacy of paclitaxel coated PTA balloons; in inhibiting restenosis of below the knee arteries (late lumen loss)
MeSH Terms: conditions — Atherosclerosis | interventions — Angioplasty, Balloon

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Placebo Comparator): Normal balloon for balloon angioplasty (Submarine, Ampherion Deep by Invatec)
  Interventions: Device: Balloon angioplasty (uncoated conventional balloon)
- 2 (Active Comparator): Paclitaxel coated balloon (same balloon like in the control group, but coated with 3 µg/mm2 Paclitaxel)
  Interventions: Device: Balloon angioplasty (conventional but coated with 3 µg/mm2 paclitaxel)

INTERVENTIONS:
Device: Balloon angioplasty (uncoated conventional balloon) — endovascular therapy
  Arms: A
Device: Balloon angioplasty (conventional but coated with 3 µg/mm2 paclitaxel) — endovascular therapy
  Arms: 2

SUMMARY:
The study will be performed as a randomized, double blind trial (in respect of the primary end point) with treatment of the stenotic lesion using uncoated PTA-catheters as control group. 114 patients will be included in the trial at about 5 study centers. Follow-up includes control angiography after 6 and 18 months and clinical follow-up examinations up to 18 months. Primary objective:

Efficacy of paclitaxel coated PTA balloons in inhibiting restenosis of below the knee arteries (late lumen loss)

Secondary objective:

Various angiographic and clinical efficacy measures, safety and tolerance of pacli-taxel coated PTA balloons in inhibiting restenosis of below the knee arteries Descriptive statistics, comparison by t-test, chi-square test for binary events 10.1 Descriptive statistics As far as applicable descriptive statistics will be applied to data and will be referring to individual changes versus baseline (predilatation or immediately postdilatation). The groups will be compared to each other testing the statistical significance of differences (p ≤ 0.05). Con-tinuous data will be expressed as mean ± standard deviation.

Categorical variables will be compared using the chi-squared test, and continuous variables will be compared using Student's t test or ANOVA analysis.

In addition to the assessment of the primary endpoint and the secondary endpoints a multi-variate analysis to investigate the influence of risk factors on the interventional outcome (interventional success, early restenosis/occlusion, LLL, stent integrity) and clinical outcomes will be performed. For this analysis the following factors will be considered: age, diabetes, neurological status (only Rutherford 5), lesion length, grade of dissection and calcification, reststenosis, number of run-off vessels, stent administration in the index lesion(s).

10.2 Estimated number of patients The primary endpoint of the study is late lumen loss (LLL) at 6 months evaluated by quantitative angiography. Because no data according this endpoint are available for both the control group and the group which will be treated with the paclitaxel coated balloon an assumption according the LLL at 6 months was made according the expectations of the principle investigator. An estimate for LLL as % of MLD in the control group is 50% and in the drug coated balloon group 30 %. The standard deviation is calculated to be 30% of LLL. A sample size of 37 patients in each group will allow the detection of a statistically significant difference (p<0.05) with 80% power. Based on the "Below study" which enrolled patients with comparable arterial lesions in Tuebingen and the data of the Basil study, it is estimated that 35% of the patients who will be enrolled in the study will not be available for follow-up investigations in order to calculate the MLD.

In order to meet a statistical endpoint a total of 114 patients will be enrolled.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 95 years,
* peripheral vascular disease, Rutherford stage 3-5, diameter stenosis ≥ 70 %, ≥ 15 -150 mm length, up to 2 vessels to be treated

Exclusion Criteria:

* Disease associated with life-expectancy less than 18 months
* Acute thrombus or aneurysm in the index limb/ vessel
* Doubts in the willingness or capability of the patient to allow follow up examination

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 114 (Estimated)
Dates: Start 2008-04; Primary Completion 2011-04 (Estimated); Study Completion 2011-04 (Estimated)

PRIMARY OUTCOMES:
Primary endpoint: Late lumen loss (LLL) of the target lesion after 6 months (assessed by DSA) | after 6 months

SECONDARY OUTCOMES:
Interventional success rate (defined as reststenosis less than 50%) | up to 18 months
Restenosis rate at 6 and 18 months (restenosis rate is defined as a diameter stenosis of ≥ 50% of reference diameter | up to 18 months
Minimum lumen diameter (MLD) at 6 months | up to 18 months
Target lesion revascularization recorded at 6, 12 and 18 months; target lesion revascularization is defined as any reintervention or artery bypass graft surgery involving the target lesion. | up to 18 months
Target vessel revascularization recorded at 6, 12 and 18 months | up to 18 months
Target limb revascularization recorded at 6, 12 and 18 months | up to 18 months
Improvement of clinical stage at 6, 12 and 18 months | up to 18 months
Change in ABI compared to pretreatment if vessels are compressible | up to 18 months
Hospitalization (extra days due to complications of the index procedure) and hospitalization between the follow-up visits due to the index leg | up to 18 months
Major amputations at the index limb | up to 18 months
Mortality | up to 18 months
LLL of stented segments at 6 months comparing the uncoated and the coated bal-loon group. | up to 18 months
Subgroup analysis; primary endpoint and TLR | up to 18 months
LLL, MLD and restenosis rate at 18 month follow-up determined by angiography | up to 18 months
Subgroup analysis neuropathy and no neuropathy according to clinical improve-ment in patients classified Rutherford 5 | up to 18 months
Clinical benefit patients Rutherford 3 vs. Rutherford 4 and 5 | up to 18 months

CONTACTS AND LOCATIONS:
Locations (5):
- Germany (5):
  - Herzzentrum Bad Krozingen, Bad Krozingen, Baden-Wurttemberg
  - University of Tuebingen, Tübingen, Baden-Wurttemberg
  - Charite Berlin, Berlin, B
  - Jüdisches Krankenhaus Berlin, Berlin, B
  - University of Rostock, Rostock, MP

REFERENCES:
- [Background] Tepe G, Zeller T, Albrecht T, Heller S, Schwarzwalder U, Beregi JP, Claussen CD, Oldenburg A, Scheller B, Speck U. Local delivery of paclitaxel to inhibit restenosis during angioplasty of the leg. N Engl J Med. 2008 Feb 14;358(7):689-99. doi: 10.1056/NEJMoa0706356. PMID 18272892